CLINICAL TRIAL: NCT06421116
Title: Validation of a Preclinical Model Based on Patient-derived Organoids for the Study of the Gut-joint Axis in Spondyloarthritis
Acronym: ORGANOSPA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6378
Record Dates: First submitted 2024-02-09; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-02

CONDITIONS: Spondyloarthritis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Spondylarthritis; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Synovial biopses and intestinal biopses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Synovial ultrasound-guided biopsy Intestinal biopsy — Patients will undergo biopsies if needed for standard-of-care follow-up and after clinical indication.

SUMMARY:
This project aims to develop and validate a model of human organoids derived from patients with Spondyloarthritis, focusing on synovial and intestinal tissues as targets of the gut-joint axis. The tissue marker profile of patient-derived organoids studied by gene expression, immunohistochemistry, and cytokine production profile will be compared with that of controls in order to test for the presence of specific biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age;
* Ability to understand and sign an informed consent form;
* Clinical indication for intestinal and/or synovial biopsy;
* Only for SpA patients group: meeting ASAS classification criteria.

Exclusion Criteria:

* Actively treated cancer;
* Severe comorbidities that, in the investigator's opinion, may affect the quality of samples for planned experimental applications;
* Only for patients undergoing ileal-colic biopsy: history of colorectal cancer disease, celiac disease;
* Only for patients undergoing a synovial biopsy: septic arthritis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients affected by Spondyloarthtitis. Controls with inflammatory or non-inflammatory conditions.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Viability assessment | 24 months
  The viability of organoids will be determined using an adenosine triphosphate (ATP) detection assay based on luminescence using a commercially available luciferase.

SECONDARY OUTCOMES:
Production of pro-inflammatory cytokines | 24 months
  The production of cytokines in the culture supernatant of organoids will be evaluated using enzyme-linked immunosorbent assay (ELISA)

OTHER OUTCOMES:
Invasion capacity assessment (synovial organoids) | 24 months
  Fibroblast-like synoviocytes (FLS) will be dispensed into a well of a Fluorobook invasion plate. The fluorescence will be measured as an index of FLS invasion capacity in the presence of a basement membrane extract.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, RM, Italy